CLINICAL TRIAL: NCT03453307
Title: The Correlation Study of the Drug Sensitivity Between Ex Vivo Model of Non-Small Cell Lung Cancer (NSCLC) Patient-Derived Organoids and Clinical Response in NSCLC Patients
Brief Title: Drug Sensitivity Correlation Between Patient-Derived Organoid Model and Clinical Response in NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: K2 Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: K2OLC-001
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: NSCLC
Keywords: Tumor Organoids; Drug Sensitivity; NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Tumor samples from surgical resection of enrolled NSCLC patients are to be collected, and subject to organoid isolation followed by ex vivo drug sensitivity test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group-1: NSCLC patients receiving chemotherapy or target therapy treatment.

SUMMARY:
This clinical study aims to evaluate the feasibility to predict clinical response of target therapy or chemotherapy drugs based on the ex vivo drug sensitivity data using patient-derived organoids.

DETAILED DESCRIPTION:
Methods - Open label single arm observatory comparison experiment

1. Enrolled patients (before or after surgery) were treated with chemotherapy or target therapy. The medication regime and treatment cycle were decided based on the clinical guideline and evidence-based medicine. This clinical study will not affect the treatment plan of the patients.
2. The resection tissue or biopsy tissue of NSCLC will be collected, and subject to ex vivo 3-D culture to establish patient-derived tumor organoid models, which will be used for drug sensitivity test.
3. The patient-derived organoid-based drug sensitivity test will be compared with clinical treatment data of chemotherapy or target therapy, followed by correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or more;
* Late stage NSCLC patients, with tumor invasion confirmed by histopathology analysis. Metastasis of axillary lymph nodes and other region lymph nodes are confirmed with histopathologic or cytopathologic analysis;
* Accessible to biopsy and/or surgery sample of metastasis and/or primitive tumor;
* No clinical evidence of other malignancy, unstable complication or uncontrolled infection;
* Life expectancy > 12 months.
* Informed and signed consent by the patient.

Exclusion Criteria:

* Not accessible to biopsy and/or surgery sample;
* Patient already enrolled in another clinical trial with another first line of chemotherapy;
* Unmeasurable locally advanced (incurable) or metastatic lesion(s), according to RECIST 1.1 criteria;
* Women who are pregnant, plan to become pregnant or are lactating during the study;
* Elevation of carcinoembryonic antigen (CEA) observed without distal metastases found;
* Have some kind of contraindications for chemotherapy and targeted therapy: cardiovascular and cerebrovascular diseases; liver and kidney function deficiency; hematological system diseases; clinician consider the patients are not suitable for chemotherapies or target therapies;
* Have other malignant tumor previously;
* Have surgical contraindications: anesthesia taboo; surgery unresectable extensive lesions;
* State of health can't finish the study;
* Patient already enrolled in another clinical trial with another anti-cancer therapy or plan to participate in other clinical study.
* No self-determination or refuse to participant.
* With unlisted exclusion criteria but are considered not suitable for the clinical study by researchers.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Metastatic NSCLC patients with axillary and other region lymph nodes metastasis. The biopsy and/or surgery tissue samples of metastatic and/or primitive tumor are accessible.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of ex vivo sensitivity test on patient derived organoid models | 12 months
  The drug sensitivity was tested on patient-derived tumor organoids, which is compared with clinical response of the chemo or target therapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Sun, Dr., Principal Investigator — K2 Oncology, Inc.
Locations (1):
- People's Hospital of Hebei Province, Shijiazhuang, Hebei, China